CLINICAL TRIAL: NCT01281319
Title: Evaluation of a Diagnostic Kit for the Detection of Serum Antibodies Anti Genital Mycoplasma in High Risk Pregnant Women
Brief Title: Evaluation of a Serology Diagnostic Kit for the Detection of Genital Mycoplasma in Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Promyco Diagnostics (Industry)
Collaborators: Soroka University Medical Center (Other)
Responsible Party: Dr Offer Erez, Soroka Medical Center
Other Study IDs: SOR510010CTIL
Record Dates: First submitted 2011-01-20; First posted 2011-01-21 (Estimated); Last update posted 2011-01-21 (Estimated); Status verified 2011-01

CONDITIONS: Genital Mycoplasma Infection; High Risk Pregnancy; Preterm Labor
Keywords: preterm labor; PROM; mycoplasma; ureaplasma; high risk pregnancy
MeSH Terms: conditions — Obstetric Labor, Premature; Mycoplasma Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cervix swab, amniotic fluid and serum samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Asymptomatic normal pregnant women
- Women with high risk pregnancy: Women at risk for preterm birth or recurrent abortions that are being followed at the high risk pregnancy unit (outpatients clinic, high risk day care center)
- Women admitted with preterm labor: Women that are admitted to the gynecology department due to pregnancy complications: preterm labor with intact membranes (PTL) or with preterm PROM.

SUMMARY:
Subclinical urogenital infections have been implicated in up to 70% of adverse pregnancy outcome, especially preterm labor and delivery. The most prevalent microorganisms involved in intrauterine infections are urogenital Mycoplasmas. Diagnosis by culturing or PCR merely detect the presence of the bacteria, pointing to colonized carriers only. There is no efficient and reliable diagnostic test to identify those subjects that have developed an infectious disease and are at risk of developing adverse pregnancy outcome.

In order to identify women at risk for developing pregnancy complications, Promyco Diagnostics has developed a proprietary, simple and non-invasive serology diagnostic kit for the detection of urogenital Mycoplasma infection.

DETAILED DESCRIPTION:
Preterm labor and delivery are the major causes of peri-natal mortality and morbidity, accounting for 9-13% of all births, and associated with over 75% of infant mortality.

Subclinical urogenital infections have been implicated in up to 70% of adverse pregnancy outcome, especially preterm labor and delivery . The most prevalent microorganisms involved in intrauterine infections are urogenital Mycoplasmas. These bacteria are frequently found in the lower genital tract of sexually active men and women and are often considered as normal flora. However, Mycoplasma can spread and colonize the internal membranes and elicit an inflammatory response in the uterus initiating the cascade of events leading to precipitous delivery. It may also cause additional pregnancy complications such as chorioamnionitis, recurrent spontaneous abortions and postpartum endometritis.

Traditional diagnostic methods, such as microbial culturing or PCR, merely detect the presence of the bacteria, pointing to colonized carriers only. There is no efficient and reliable diagnostic test to identify those subjects that have developed an infectious disease and are at risk of developing adverse pregnancy outcome.

Studies show that colonization of the cervix or amniotic fluid alone cannot accurately predict pregnancy complications. In contrast, identification of antibodies to Mycoplasma in colonized women predicted an outstanding 85-90% of low birth weight or preterm delivery respectively.

In order to identify women at risk for developing pregnancy complications, Promyco Diagnostics has developed a proprietary, simple and non-invasive serology diagnostic kit for the detection of urogenital Mycoplasma infection.

ELIGIBILITY:
Inclusion Criteria:

1. Women who are 18 years of age or older.
2. Normal pregnancy at first trimester, or
3. Women admitted with PTL, defined as the presence of regular uterine contractions associated with progressive effacement and dilatation of the uterine cervix, or
4. Women admitted with PROM, defined as rupture of the chorioamniotic membranes before the onset of labor and diagnosed by sterile speculum examination confirming pooling of amniotic fluid in the vagina, positive nitrazine test or incase of diagnostic amniocentesis leakage of indigocarmine through the uterine cervix, or
5. Women admitted with chorioamnionitis, an inflammation of the fetal membranes (amnion and chorion), or
6. Past pregnancy complications, including recurrent abortions, stillbirth, fetal loss, history of spontaneous preterm labor and/or delivery, or
7. Recurrent abortions

Exclusion Criteria:

1. High risk pregnancy due to: gestional diabetes, preeclampsia, small for gestational age fetus.
2. Multiple gestation.
3. Pre-existing chronic illness - high blood pressure, heart disease, diabetes, lupus, asthma, a seizure disorder, or another longstanding medical problem.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Normal and high risk pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the novel serology kit | December 2011
  Assess the efficacy of the novel serology diagnostic kit for the detection of anti-urogenital Mycoplasma antibodies in the maternal serum
Antibody titer according to gestational age | December 2011
  Determine the changes in antibody titer according to gestational age both in normal and complicated pregnancies.
Correlation between culture and serology | December 2011
  Determine the correlation between the antibody titer and the presence of urogenital Mycoplasma in cervix and/or amniotic fluid cultures of high risk pregnant women.
Correlation between antibody titer and pregnancy outcome | Dec 2012
  Determine the correlation between maternal serum anti urogenital Mycoplasma antibody titer and pregnancy outcome in patients at risk for spontaneous preterm birth.

CONTACTS AND LOCATIONS:
Overall Officials: Offer Erez, MD, Principal Investigator — Soroka University Medical Center
Locations (1):
- Soroka University Medical Center, Beersheba, Israel

REFERENCES:
- [Background] Horowitz S, Mazor M, Horowitz J, Porath A, Glezerman M. Antibodies to Ureaplasma urealyticum in women with intraamniotic infection and adverse pregnancy outcome. Acta Obstet Gynecol Scand. 1995 Feb;74(2):132-6. doi: 10.3109/00016349509008922. PMID 7900509
- [Background] Cassell GH, Davis JK, Waites KB, Rudd PT, Talkington D, Crouse D, Horowitz SA. Pathogenesis and significance of urogenital mycoplasmal infections. Adv Exp Med Biol. 1987;224:93-115. doi: 10.1007/978-1-4684-8932-3_10. PMID 3329816
- [Background] Horowitz S, Mazor M, Romero R, Horowitz J, Glezerman M. Infection of the amniotic cavity with Ureaplasma urealyticum in the midtrimester of pregnancy. J Reprod Med. 1995 May;40(5):375-9. PMID 7608879